CLINICAL TRIAL: NCT04991064
Title: Retention of Maxillary Complete Dentures Modified With Titanium Dioxide Nanoparticles: A Randomized Crossover Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Gamal Ismail Mohamed, Dr, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 38912240102212
Record Dates: First submitted 2021-07-17; First posted 2021-08-05 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Denture Retention; Complete Dentures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB arm (Other): participants allocated to this arm receive treatment A first, followed by treatment B.
  Interventions: Other: Complete denture base modified by Titanium dioxide nanoparticles.
- BA arm (Other): participants allocated to this arm receive treatment B first, followed by treatment A.
  Interventions: Other: Complete denture base modified by Titanium dioxide nanoparticles.

INTERVENTIONS:
Other: Complete denture base modified by Titanium dioxide nanoparticles. — Titanium dioxide nanoparticles will be mixed with resin powder of the denture base before mixing the powder and liquid of the heat cure denture base material.

SUMMARY:
This study investigates the effect of the addition of titanium dioxide nanoparticles to denture base materials on their retention compared to that of the unmodified denture base materials.

DETAILED DESCRIPTION:
All patients will be randomly allocated to two equal groups either with the protocol I or II (5 in each group) with an allocation ratio of 1:1 through a computer-generated sequence by a spreadsheet (Excel, Microsoft Office 2010; Microsoft Corp). The group with the protocol I will use the modified dentures with titanium dioxide nanoparticles (TiO2NP) during the first month, followed by no use of the first denture and the use of their old relined dentures instead for 1 month (washout), and then the use of the unmodified dentures for 1 month; the group with the protocol II will use the unmodified dentures during the first month, followed by no use of the first denture and the use of their old relined dentures instead for 1 month (washout), and then the use of the modified dentures TiO2NP for 1 month. Assessment of retention will be done immediately and 1 month after denture insertion.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring new removable complete dentures, with class I edentulous arches based on the American College of Prosthodontists (ACP) classification15, with an average age of 45-55 years old, with healthy temporomandibular joint, being without systemic disease that could affect the neuromuscular control or salivary flow

Exclusion Criteria:

* Patients with ACP Class II, III, or IV, and xerostomia.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the change in the retention within each type of complete denture. | Assessment will be done Immediately and 1 month after denture insertion within each type of denture.
  It is measured in Newton.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: No
Only the co-author has the IPD. He is responsible to store it in an inaccessible place for anyone.